CLINICAL TRIAL: NCT03503227
Title: The Value of Addition of Prednisolone to Acetylsalicylic Acid Prior to Embryo Transfer in Patients With First ICSI Cycles: A Randomized Controlled Trial
Brief Title: The Value of Prednisolone With Aspirin Before Embryo Transfer in Intracytoplasmic Sperm Injection (ICSI) Cycles
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amira S Dieb, Ob/Gyn Lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1199012
Record Dates: First submitted 2018-04-02; First posted 2018-04-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Active Comparator): Patients will receive daily oral low dose Acetylsalicylic acid (75 mg) starting day 20 of the previous cycle withGonadotrophin releasing hormone agonist (GnRH agonist)
  Interventions: Drug: Acetyl Salicylic acid
- Aspirin and prednisolone (Active Comparator): Patients will receive daily oral low dose Acetylsalicylic acid (75 mg) and Low dose prednisolone (10 mg/day) starting day 20 of the previous cycle withGonadotrophin releasing hormone agonist (GnRH agonist).
  Interventions: Drug: prednisolone; Drug: Acetyl Salicylic acid

INTERVENTIONS:
Drug: prednisolone — daily oral low dose prednisolone (10 mg/day) :a glucocorticoid
  Arms: Aspirin and prednisolone
Drug: Acetyl Salicylic acid — daily oral low dose Acetylsalicylic acid (75 mg) : Antiplatelet agent

SUMMARY:
This study is a prospective, double-blind, randomized controlled trial . It includes 250 infertile patients scheduled for ICSI cycle. The patients will be randomly allocated into two equal groups; daily oral low dose Acetylsalicylic acid and group B patients will receive daily oral low dose Acetylsalicylic acid and Low dose prednisolone. All 250 participants undergo similar ICSI cycles. Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include number of oocytes retrieved, fertilization rate, number of embryos, embryo quality, chemical pregnancy rate, twins rate and miscarriage rate per cycle.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled trial. Patients undergoing ICSI for their first cycle are enrolled in this study. Participants are then randomized into two groups ; group A patients will receive daily oral low dose Acetylsalicylic acid (75 mg) and group B patients will receive daily oral low dose Acetylsalicylic acid (75 mg) and Low dose prednisolone (10 mg/day).

Randomization will be done by withdrawing closed envelopes for each patient .

Inclusion criteria:

Women in reproductive age diagnosed with infertility for ICSI, female age (18- <40 years, normal serum hormonal profile on day 3 of the cycle [including estradiol (E2), follicle stimulating hormone (FSH), Luteinizing hormone (LH), prolactin, thyroid stimulating hormone, normal uterine cavity diagnosed at hysteroscopy.

Exclusion criteria:

* Women with platelet dysfunction, thrombocytopenia, gastrointestinal ulcers, recurrent gastritis, Acetylsalicylic acid hypersensitivity, patients on corticosteroids will be excluded from the study.
* Also women with known cause for recurrent miscarriage: antiphospholipid syndrome, abnormal thyroid function tests, parental balanced translocation or uterine anomaly (known subseptate uterus or cervical weakness diagnosed at hysteroscopy).
* Contraindications to steroid therapy: hypertension, diabetes, mental health problems or obesity with Body mass index (BMI) >35
* Decline consent to randomization

Methodology in details:

All patients will be subjected to the following:

* -Informed consent after explaining the aim of the study, procedure and possible hazards.
* -History taking includes full obstetric history, medical and surgical history and demographic distribution.
* Full physical examination. -
* -Ultrasound examination (2D): Transvaginal sonography (TVS) is done on day 2 to 5 to assess antral follicle count (AFC), uterus and adnexa .
* -Each group will start intake of Acetyl-Salicylic Acid (ASA) or ASA with Prednisolone on day 19th - 20th of the previous cycle and continue until confirmation of pregnancy by detection of fetal heart activity on ultrasound.
* -Long protocol steps:

  * Start from day 19th - 20th by GnRH agonist ;Triptorelin 0.1mg subcutaneous (Decapeptyl, Ferring). -1st visit : after 2 weeks of start of GnRH agonist or day 2 of cycle, we confirm down regulation by a serum level of E2to be <50 pg/ml, endometrial thickness <5mm, no ovarian cyst by ultrasound. Then we add Gonadotropins as Intramuscular (I.M.) injections of 150-300 I.U. of highly purified Human Menopausal Gonadotropins daily (Merional, 75 I.U. /vial, IBSA). The dose is adjusted according to the age, BMI, AFC, serum levels of anti-mullerian hormone (AMH), follicle stimulating hormone (FSH) and ovarian response.
  * 2nd visit : on 6th - 7 th days of Gonadotrophins and then every other day to do folliculometry by TVS and E2 level in serum.
  * We do trigger by Human Chorionic Gonadotrophin (HCG)10000 IU I.M.(Pregnyl, Organon) when at least 3 follicles reach 18mm in mean diameter or more and E2 level is less than 2500 pg/ml. Ovum pickup is done 34 hours after HCG injection and embryo transfer using Wallace catheter on day 2 to 3.
* -Luteal support: Natural Progesterone 400 mg 1x2, Folic acid once daily, Amoxicillin-Clavulanic Acid 1gm 1x2x7 ,Progesterone 100mg I.M. daily for 10 days, Acetylsalicylic Acid once daily
* -Quantitative ß- HCG in serum after 14 days of embryo transfer. -TVS to detect clinical pregnancy at 6-7 weeks of gestation.

Primary outcome:

The primary outcome is clinical pregnancy rate per cycle.

Secondary outcome:

Secondary outcome measures are number of oocytes retrieved, fertilization rate, number of embryos, embryo quality, chemical pregnancy rate, twins rate and miscarriage rate per cycle.

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive age diagnosed with infertility for IVF/ICSI, female age (18- <40 years, normal serum hormonal profile on day 3 of the cycle [including estradiol (E2), FSH, LH, prolactin, thyroid stimulating hormone, normal uterine cavity diagnosed at hysteroscopy.

Exclusion Criteria:

* Women with platelet dysfunction, thrombocytopenia, gastrointestinal ulcers, recurrent gastritis, Acetylsalicylic acid hypersensitivity, patients on corticosteroids will be excluded from the study.
* Also women with known cause for recurrent miscarriage: antiphospholipid syndrome (positive anticardiolipin antibody or lupus anticoagulant on 2 separate occasions at least 6 weeks apart), thrombophilia (factor V Leiden mutation, activated protein C resistance (APCR) resistance, protein C or S deficiency, prothrombin gene mutation, antithrombin III deficiency), abnormal thyroid function tests, parental balanced translocation or uterine anomaly (known subseptate uterus or cervical weakness diagnosed at hysteroscopy).
* Contraindications to steroid therapy: hypertension, diabetes, mental health problems or obesity with BMI >35
* Decline consent to randomization

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per cycle. | 7 weeks
  Detection of gestational sac , embryo pole and fetal pulsations by transvaginal ultrasound

SECONDARY OUTCOMES:
number of oocytes retrieved per cycle. | 3 weeks
  number of oocytes retrieved during ovum pickup per cycle.
fertilization rate per cycle. | 3weeks
  The number of oocytes fertilized by intracytoplasmic sperm injection per cycle.
number of embryos per cycle. | 3weeks
  number of embryos of any grade ( first, second, third or fourth grade) per cycle
embryo quality per cycle. | 3weeks
  embryo quality by grade ( first, second, third or fourth) per cycle.
chemical pregnancy rate per cycle. | 5 weeks
  Positive beta hCG in serum per cycle.
twins rate per cycle. | 9 weeks
  Detection of 2 gestational sacs with positive fetal poles and pulsations per cycle.
miscarriage rate per cycle. | 16 weeks
  Early pregnancy loss per cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Amira S Dieb, MD, Principal Investigator — KasrAlainiH
Locations (1):
- KasralainiH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No